CLINICAL TRIAL: NCT01844414
Title: Health Promotion Coaching/Vaccine for Homeless Parolees
Brief Title: UCLA-Amity Parolee Health Promotion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adeline Nyamathi, PhD, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10000358
Record Dates: First submitted 2013-03-21; First posted 2013-05-01 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis B; Hepatitis C; HIV; Drug Addiction
Keywords: Homeless Men; Parolees; Hepatitis B; Hepatitis C; HIV; Community Drug Treatment; Recidivism
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Substance-Related Disorders; Recidivism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Parolee Comprehensive Care + Phone Coach (Experimental): PCPC Intervention: Eight specialized nurse case managed hepatitis education sessions, the Hepatitis A/B vaccine series and coach-facilitated mentoring.
  Interventions: Behavioral: Parolee Comprehensive Care + Phone Coach
- Parolee Brief HBV program + Phone Coach (Experimental): PBPC Intervention: Eight twenty minute hepatitis education sessions, coach facilitated mentoring and the Hepatitis A/B vaccine series.
  Interventions: Behavioral: Parolee Brief HBV Program + Phone Coach
- Usual Care Group (Active Comparator): UC Control Group: One brief general health information program, one-on-one coaching and the Hepatitis A/B vaccine.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Parolee Comprehensive Care + Phone Coach — A nurse case managed and specialized hepatitis education program with the hepatitis A/B (HAV/HBV) vaccination series (to all eligible) and coach-facilitated mentoring (mostly by cell-phone).
  Other Names: PCPC
  Arms: Parolee Comprehensive Care + Phone Coach
Behavioral: Parolee Brief HBV Program + Phone Coach — A brief hepatitis/HIV education program with the Hepatitis A/B vaccine series and coach-facilitated mentoring.
  Other Names: PBPC
  Arms: Parolee Brief HBV program + Phone Coach
Behavioral: Usual Care Group — Control Group: A brief general health information program with one-on-one coaching and the Hepatitis A/B vaccine
  Other Names: UC
  Arms: Usual Care Group

SUMMARY:
The purpose of this study is to conduct a prospective, three-group study that randomly assigns 700 parolees, in a community residential drug treatment program, to enter one of three groups: 1) a PCPC (Parolee Comprehensive Care + Phone Coaching Program), which includes nurse case management and specialized hepatitis education sessions and the hepatitis A/B (HAV/HBV) vaccination series (to all eligible) and coach-facilitated mentoring (mostly by cell-phone); 2) a Parolee Brief Hepatitis Education + HBV vaccination + Phone Coaching (PBCP) Program, which includes brief hepatitis/HIV education, HAV/HBV vaccination and coach-facilitated mentoring; or 3) a Usual Care (UC) control program, which includes brief general health information, one-on-one coaching and the HAV/HBV vaccine.

DETAILED DESCRIPTION:
Homeless parolees pose a particular challenge for successful reentry into the community as they have underlying mental health issues combined with substance use and abuse and must contend with unstable housing situations, disorganized lives, unemployment, and limited access to health care and social services. Generally about 50% of all parolees scheduled to enroll in community-based drug treatment fail to enroll and less than 10% of enrollees actually complete treatment. Not surprisingly, about two-thirds of all individuals on parole are rearrested and return to custody within three years of release from prison. Recent data also revealed homeless persons who were least likely to complete a Hepatitis A/B (HAV/HBV) vaccine series were young (< 40) men who had been discharged from prison. Therefore, it is critical to engage paroled adults in comprehensive intervention programs that not only protect them from hepatitis B, but also reduce risky behavior, promote access to health care, social and employment services, and enable positive coping and communication skills.

Building upon advice from community partners who have successfully treated parolees and the research team's experience with hepatitis vaccination work, this study is designed to conduct a prospective, three-group study that randomly assigns 700 ready-for-discharge parolees, scheduled to enter a community residential drug treatment program, to enter one of three groups: 1) a PCPC (Parolee Comprehensive Care + Phone Coaching Program), which includes nurse case management and specialized hepatitis education sessions and referrals, the HAV/HBV vaccination series (to all eligible) and coach-facilitated mentoring (mostly by cell-phone); 2) a Parolee Brief Hepatitis Education + HBV vaccination + Phone Coaching (PBCP) Program, which includes brief hepatitis/HIV education, the HAV/HBV vaccination and coach-facilitated mentoring; or 3) a Usual Care (UC) control program, which includes brief general health information, and the HAV/HBV vaccine. This study will advance the research team's knowledge about drug treatment and HBV vaccine completion and recidivism among homeless parolees. Findings from this study can inform targeted interventions and lay the groundwork for health policy decisions that may impact hepatitis and HIV risk reduction and recidivism in this group who are a reservoir for these viruses in the general population, and are returning to prison at unprecedented numbers.

ELIGIBILITY:
Inclusion Criteria:

1. Parolees enrolled in Amity's Amistad's program;
2. Age 18-60;
3. Discharged from prison or jail within the last six months;
4. History of drug use 12 months prior to most recent incarceration;
5. Previously homeless prior to most recent incarceration; and
6. Willing to provide informed consent

Exclusion Criteria:

1. Monolingual speakers of languages other than English; and
2. Persons judged to be cognitively impaired by the research staff.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2010-02; Primary Completion 2014-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 5 years
  ● Number of re-incarcerations
Primary Outcome Measure | 5 years
  ● Completion of the Hepatitis A/B vaccine (for HBV negative participants);
Primary Outcome Measure | 5 years
  ● Completion of six months of a community-based residential drug treatment program;

SECONDARY OUTCOMES:
Secondary Outcome Measure | 5 years
  Reduction in drug and alcohol use and sexual risk behaviors;
Secondary Outcome Measure | 5 years
  Number of visits to health care or social service providers;
Secondary Outcome Measure | 5 years
  Improved knowledge of Hepatitis/HIV and communication skills between 6 and 12 months or over the one-year study period;
Secondary Outcome Measure | 5 years
  Cost Effectiveness of each of the three programs

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Nyamathi, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Amistad de Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Nyamathi A, Marlow E, Zhang S, Hall E, Farabee D, Marfisee M, Khalilifard F, Faucette M, Leake B. Correlates of serious violent crime for recently released parolees with a history of homelessness. Violence Vict. 2012;27(5):793-810. doi: 10.1891/0886-6708.27.5.793. PMID 23155727
- [Result] Nyamathi A, Leake B, Albarran C, Zhang S, Hall E, Farabee D, Marlow E, Marfisee M, Khalilifard F, Faucette M. Correlates of depressive symptoms among homeless men on parole. Issues Ment Health Nurs. 2011;32(8):501-11. doi: 10.3109/01612840.2011.569111. PMID 21767252
- [Derived] Nyamathi AM, Zhang SX, Wall S, Hall EA, Salem BE, Farabee D, Faucette M, Yadav K. Drug Use and Multiple Sex Partners Among Homeless Ex-Offenders: Secondary Findings From an Experimental Study. Nurs Res. 2016 May-Jun;65(3):179-90. doi: 10.1097/NNR.0000000000000150. PMID 27124254
- [Derived] Nyamathi A, Salem BE, Zhang S, Farabee D, Hall B, Khalilifard F, Leake B. Nursing case management, peer coaching, and hepatitis a and B vaccine completion among homeless men recently released on parole: randomized clinical trial. Nurs Res. 2015 May-Jun;64(3):177-89. doi: 10.1097/NNR.0000000000000083. PMID 25932697